CLINICAL TRIAL: NCT00287313
Title: Use of Daily Vitamin K Supplementation in Patients on Warfarin With a History of Frequent Dose Changes or Variable INRs
Brief Title: Daily Vitamin K in Patients on Warfarin With Unstable INRs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Stephan Moll, MD, University of North Carolina at Chapel Hill
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-MED-491
Record Dates: First submitted 2006-02-03; First posted 2006-02-06 (Estimated); Last update posted 2010-01-12 (Estimated); Status verified 2010-01

CONDITIONS: Anticoagulants; Warfarin
Keywords: Unstable INRs; Warfarin; Vitamin K
MeSH Terms: interventions — Vitamin K

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Vitamin K

SUMMARY:
The purpose of this study is to determine if daily Vitamin K supplementation stabilizes INRs in patients taking warfarin with a history of frequent dose changes or variable INRs.

DETAILED DESCRIPTION:
Consistent daily Vitamin K intake may contribute to the stabilization of INR values in patients with unstable INRs on warfarin therapy. Subjects with unstable INRs will be identified from the existing patient records of the UNC Anticoagulation Clinics. Eligible subjects will sign an informed consent form and will receive a point-of-care (POC) INR monitoring device. They will undergo 9 weeks of home INR monitoring via the POC device (with monthly clinic follow-up). They will subsequently be provided with 500 mcg Vitamin K tablets to be taken once daily. Weekly POC INR monitoring with monthly clinic follow-up will continue for an additional 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patient of UNC Anticoagulation Clinic with INR target of 2.0-3.0 and at least 9 months on uninterrupted warfarin
* Unstable INRs for the past 6 months, defined as a minimum number of warfarin dose changes of 3
* Patient demonstration of proper POC device technique on 2 measurements during one teaching session with investigator
* Age greater than or equal to 18 years

Exclusion Criteria:

* Stroke or TIA within the previous 12 months
* VTE within the last 3 months
* Antiphospholipid antibody syndrome
* Pregnant patients, since warfarin is contraindicated during pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2005-10; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Number of warfarin adjustments required in each phase
Time in therapeutic, sub-, and supra-therapeutic range
Variance/SD of INRs for each patient
Adherence assessed by pill counts and pharmacy record review
Thrombotic/bleeding episodes

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Moll, M.D., Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States